CLINICAL TRIAL: NCT00734708
Title: Phase 3 Clinical Trial of Periodontal Tissue Regeneration Using Fibroblast Growth Factor-2(Trafermin)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KCB-1D-03
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Periodontitis; Alveolar Bone Loss; Periodontal Attachment Loss
MeSH Terms: conditions — Periodontitis; Alveolar Bone Loss; Periodontal Attachment Loss | interventions — trafermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): positive drug (0.3% Trafermin contained)
  Interventions: Drug: Trafermin (genetical recombination)
- P (Placebo Comparator): control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trafermin (genetical recombination) — Administered to the bone defect during flap operation
  Other Names: KCB-1D
  Arms: A
Drug: Placebo — Control
  Arms: P

SUMMARY:
This study aims to verify the effectiveness of Trafermin (recombinant human basic fibroblast growth factor) in stimulating regeneration of periodontal tissue lost by periodontitis and to evaluate the safety of such stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Probing pocket depth 4mm or deeper
* Vertical intrabony defect 3 mm or deeper from radiographs at baseline
* Mobility of tooth 2 degree or less

Exclusion Criteria:

* Using an investigational drug within the past 24 months
* Coexisting malignant tumour or history of the same
* Coexisting diabetes (HbA1C 6.5% or more)
* Taking bisphosphonates
* Coexisting gingival overgrowth or history of the same

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
rate of increase in alveolar bone height | 36 weeks after administration
clinical attachment level regained | 36 weeks after administration

SECONDARY OUTCOMES:
time course of increase rate in alveolar bone height | within 36 weeks after administration
time course of clinical attachment level regained | within 36 weeks after administration
time course change of periodontal tissue inspection values | within 36 weeks after administration
occurrence and level of adverse reaction | within 36 weeks after administration
serum anti-Trafermin antibody level | within 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chikara Ieda, Study Director — Kaken Pharmaceutical Co., Ltd.
Locations (21):
- Japan (21):
  - Kaken Investigational Site, Nagoya, Aichi-ken
  - Kaken Investigational Site, Matsudo, Chiba
  - Kaken Investigational Site, Fukuoka, Fukuoka
  - Kaken Investigational Site, Kitakyushu, Fukuoka
  - Kaken Investigational Site, Hiroshima, Hiroshima
  - Kaken Investigational Site, Ishikari-Tobetsu, Hokkaido
  - Kaken Investigational Site, Sapporo, Hokkaido
  - Kaken Investigational Site, Morioka, Iwate
  - Kaken Investigational Site, Kagoshima, Kagoshima-ken
  - Kaken Investigational Site, Machida, Kanagawa
  - Kaken Investigational Site, Yokohama, Kanagawa
  - Kaken Investigational Site, Sendai, Miyagi
  - Kaken Investigational Site, Nagasaki, Nagasaki
  - Kaken Investigational Site, Niigata, Niigata
  - Kaken Investigational Site, Okayama, Okayama-ken
  - Kaken Investigational Site, Suita, Osaka
  - Kaken Investigational Site, Tokushima, Tokushima
  - Kaken Investigational Site, Bunkyo-ku, Tokyo
  - Kaken Investigational Site, Chiyoda-ku, Tokyo
  - Kaken Investigational Site, Ōta-ku, Tokyo
  - Kaken Investigational Site, Sinjyuku-ku, Tokyo

REFERENCES:
- [Background] Kitamura M, Nakashima K, Kowashi Y, Fujii T, Shimauchi H, Sasano T, Furuuchi T, Fukuda M, Noguchi T, Shibutani T, Iwayama Y, Takashiba S, Kurihara H, Ninomiya M, Kido J, Nagata T, Hamachi T, Maeda K, Hara Y, Izumi Y, Hirofuji T, Imai E, Omae M, Watanuki M, Murakami S. Periodontal tissue regeneration using fibroblast growth factor-2: randomized controlled phase II clinical trial. PLoS One. 2008 Jul 2;3(7):e2611. doi: 10.1371/journal.pone.0002611. PMID 18596969